CLINICAL TRIAL: NCT06310161
Title: Bright Light Therapy to Treat Fatigue in End Stage Kidney Disease
Brief Title: Light Therapy in End Stage Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 855161
Record Dates: First submitted 2024-01-02; First posted 2024-03-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright Light (Experimental): Light therapy will be delivered by the Re-Timer glasses for 60 minutes during dialysis sessions.
  Interventions: Device: Bright light
- Dim Light (Placebo Comparator): Dim light therapy will be delivered by the Re-Timer glasses for 60 minutes during dialysis sessions.
  Interventions: Device: Dim Light

INTERVENTIONS:
Device: Bright light — Bright light treatment will consist of using the Re-timer device 3 times per week during dialysis sessions for 4 weeks. The Re-timer is worn like a pair of glasses and contains light emitting diodes mounted on the lower portion of the frame. The Re-timer emits blue-green 500 nm light with an intensity of ~500 lux lm/m2. Participants will be instructed to use the device for 60 minutes at the beginning of each dialysis session.
  Other Names: Re-Timer
  Arms: Bright Light
Device: Dim Light — Dim light treatment will use non-light emitting glasses that look identical to Re-Timer for 4 weeks at each dialysis session following baseline assessments. Participants will use the device for 60 minutes at the beginning of their dialysis session.
  Other Names: Re-Timer
  Arms: Dim Light

SUMMARY:
The goal of this clinical trial is to test light therapy in patients with end stage kidney disease who are receiving hemodialysis. The main aim is to determine if light therapy decreases fatigue severity. Participants will receive light therapy using special glasses for one hour during the dialysis sessions for four weeks of treatment.

DETAILED DESCRIPTION:
In a single site, 2-arm (Bright Light Therapy group; Dim Light Group), parallel, randomized controlled trial we will enroll 60 subjects (n=30 per group) to assess the effects of Bright Light Therapy compared to Dim Light Therapy in subjects with end stage kidney disease who are receiving hemodialysis to treat fatigue.

* To compare the effects of bright light therapy to dim light therapy on fatigue severity.
* To explore the effects of bright light therapy to dim light therapy on salivary cortisol.
* To compare the effects of bright light therapy to dim light therapy on insomnia, depression and quality of life.
* To test the effects on bright light therapy to dim light therapy on physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study mandated procedure
2. Male and female participants ≥ 18 years of age
3. Diagnosis end stage kidney disease with hemodialysis 3 times/week for at least 1 month
4. Fatigue Severity Scale (FSS) > 9 at enrollment
5. Home refrigerator for salivary cortisol storage

Exclusion Criteria

1. Eye disorders: cataracts, glaucoma, retinal disorders (e.g. macular degeneration)
2. Participants with photosensitivity (e.g. epilepsy)
3. Hospitalized or acutely ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 4 weeks
  Measures how bad or severe a person's fatigue is. Score range from 9-63; higher scores indicate increased fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Ann Matura, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No